CLINICAL TRIAL: NCT01903616
Title: A Longitudinal Study of Movement and Participation in Life Activities of Young Children With Cerebral Palsy in Taiwan
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NSC 98-2314-B-182-006-MY3
Record Dates: First submitted 2013-07-17; First posted 2013-07-19 (Estimated); Last update posted 2020-08-24 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study investigates the longitudinal course of developmental patterns in movement and participation in life activities (MPLA) of young children with cerebral palsy (CP) in Taiwan. Additionally, the predictors in the initial stage in determining the final developmental patterns in movement and participation in life activities MPLA of these children will be identified.

DETAILED DESCRIPTION:
Most researches investigated the longitudinal study of functions in adolescent or adult with CP, however, few researches investigate these functions in children with CP. Knowledge of these developmental patterns in movement and participation in life activities MPLA may be helpful in understanding, anticipating, and managing the problems of these children. We hypothesize that the course of developmental patterns in MPLA of young children with CP evolves with their age. This study investigates the longitudinal course of developmental patterns in MPLA of young children with CP in Taiwan. This study includes a validity and reliability study and a prospective longitudinal study of young children with CP over one-year. This study will be executed in 4 years and a validity and reliability study in the first year.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CP

Exclusion Criteria:

* presence of a progressive neurological disorder or a severe concurrent illness or disease not typically associated with CP, such as traumatic brain injury or active pneumonia

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with cerebral palsy
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2009-07; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change of speech and acoustic variables in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of speech and acoustic variables

SECONDARY OUTCOMES:
Change of range of motion (ROM) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of ROM
Change of Pediatric Berg Balance Scale (PBS) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of PBS
Change of spinal Alignment and Range of Motion Measure(SARROM) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of SARROM
Change of modified ashworth scale(MAS) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of MAS
Change of cerebral palsy quality of life (CPQOL) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of CPQOL
Change of TNO-AZL Preschool children Quality of Life (TAPQOL)in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of TAPQOL
Change of Children Assessment of Participation and Enjoyment (CAPE) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of CAPE
Change of Gross motor function measure (GMFM) in 6, 12 and 24 months | baseline, 6m, 12m, 24 m
  Measurement of GMFM

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Ling Chen, MD,PhD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No